CLINICAL TRIAL: NCT06438549
Title: Integrating CHWs Into Prenatal Care for Maternal Smoking Cessation: A Pilot Feasibility Study
Brief Title: Integrating CHWs Into Prenatal Care for Maternal Smoking Cessation
Acronym: SFHOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: University of California, San Francisco (Other); Riverside University Health System Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5220112; T32KT4784 (Other Grant/Funding Number: Tobacco-related Disease Research Program (TRDRP))
Record Dates: First submitted 2024-04-18; First posted 2024-06-03 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Tobacco Use; Tobacco Use Cessation; Tobacco Use in Childbirth
Keywords: prevention; treatment; disparities and social inequality; tobacco use cessation; community health worker; pregnant smokers
MeSH Terms: conditions — Tobacco Use; Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: The model compares the integration of CHW Home visits into healthcare provider-directed clinical care and a schedule of CHW home visits to provide behavioral smoking cessation for pregnant people and adult household members before, during, and after a quit date vs Standard of Care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated HCP-CHW Intervention Arm (Experimental): CHW visit with brief tobacco cessation intervention.
  Interventions: Behavioral: HCP-CHW Integration into Prenatal Care for Smoking Cessation
- Control arm (Other): Standard of Care
  Interventions: Other: Control Arm

INTERVENTIONS:
Behavioral: HCP-CHW Integration into Prenatal Care for Smoking Cessation — CHWs will be integrated into primary care, and subjects will receive CHW home visits (up to 8) that will provide brief behavioral smoking cessation interventions before, during, and after a quit date. This brief behavioral intervention will include watching a video and reviewing self-help materials.
  Arms: Integrated HCP-CHW Intervention Arm
Other: Control Arm — Standard of Care which provides referrals to community-based smoking cessation resources.
  Arms: Control arm

SUMMARY:
This develops a novel behavioral tobacco cessation program for pregnant smokers in San Bernardino County.

DETAILED DESCRIPTION:
This study seeks to address the disparities in the maternal smoking cessation outcomes of previous research by developing an innovative maternal tobacco cessation program that expands the outreach by integrating home visits by community health workers (CHW) into the prenatal healthcare model. The overall aim is to conduct a pilot randomized control trial to test the feasibility, acceptability, and efficacy of a Healthcare Provider-Community Health Worker (HCP-CHW) intervention model that expands outreach by adding eight home visits by CHWs to provide tobacco cessation support services before and after the quit date.

ELIGIBILITY:
Inclusion Criteria:

* < 24 weeks pregnant
* age > 18 years,
* current smokers (100 cigarettes in their lifetime and >3 cigarettes per day in the last 7 days; including poly-tobacco use, combining cigarettes with non-combustible products) confirmed by expired carbon monoxide (CO)
* willing to quit smoking and set a quit date in the next 2 weeks upon enrolling
* enrolled in prenatal care at Loma Linda University Health (LLUH) or Riverside University Health System (RUHS)

Exclusion Criteria:

* severe mental health problems that prevent informed consent and/or CHW intervention
* women who were on Nicotine Replacement Therapy (NRT) or enrolled in a cessation program within 30 days
* unwillingness to participate in audio-recorded key informant interviews or focus groups

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Self-Report Tobacco Abstinence | Change between baseline enrollment and 1 month postpartum visit, typically ten months
  The 7 Day Point Prevalence Abstinence (PPA) questionnaire will be administered to subjects to assess the following: Tobacco use within past seven days

SECONDARY OUTCOMES:
Carbon Monoxide Level | Change between baseline and 1 month postpartum visit, typically ten months
  Breathalyzer test will be administered to subjects to determine CO level. Subjects will then be classified per CO level as:
  Nonsmoker = 0 to 3 Borderline = 4 to 6 Smoker = 7 and above Smoker Low Addiction = 7 to 10 Smoker Moderate Addiction = 11 to 15 Smoker Heavily Addicted = 16 to 25 Smoker Very heavily Addicted = 26+
Arm 1 Satisfaction with CHW visit | Baseline; during the intervention; through study completion, an average of 10 months.
  The acceptability of the intervention will be assessed using composite Likert scale measures of process outcomes such as 1) overall patient satisfaction, 2) increasing patient motivation and confidence, and 3) willingness to recommend the program to others. Likert scale interpretations for overall satisfaction: 1=Very Dissatisfied; 2=Dissatisfied; 3=Neutral; 4=Satisfied; 5=Very Satisfied. Likert scale interpretation for patient motivation and confidence: 1=Strongly Disagree (The intervention did not increase motivation/confidence at all); 2=Disagree; 3=Neutral; 4=Agree; 5=Strongly Agree (The intervention significantly increased motivation/confidence). Likert scale interpretation for Willingness to Recommend the Program to Others: 1=Not at all likely; 2=Unlikely; 3=Neutral; 4=Likely; 5=Very Likely.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Berit Petersen, PhD, Principal Investigator — Loma Linda University
Locations (2):
- United States (2):
  - Loma Linda University Medical Center, Loma Linda, California
  - Riverside University Health Systems, Moreno Valley, California

REFERENCES:
- See also: Study website — https://smokefreehope.org/